CLINICAL TRIAL: NCT03914105
Title: Central Neuromodulation of Pain Through Music in Healthy Subjects (DOUMU1)
Brief Title: Central Neuromodulation of Pain Through Music in Healthy Subjects
Acronym: DOUMU1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DOUMU1 (29BRC19.0039)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without music (Active Comparator): Test without music
  Interventions: Procedure: Without music
- With music (Experimental)
  Interventions: Procedure: With music

INTERVENTIONS:
Procedure: Without music — The starting condition will be "without music": the subjects, after a rest period of 10 minutes, will perform a test of induced pain for 6 minutes. There will be no music for the duration.
  Arms: Without music
Procedure: With music — The starting condition will be "with music": the subjects, after a rest period of 10 minutes, will perform a test of induced pain for 6 minutes. There will be music for the duration.
  Arms: With music

SUMMARY:
The present research aims to study the neuromodulatory effect of music on the sensory component of pain. The activation of pain control systems, through music, would pave the way for rehabilitation prospects for patients with a deficit of these controls.

DETAILED DESCRIPTION:
Pain is a multidimensional, complex and universal phenomenon that would be faced by almost one in two European adults. To meet the needs in terms of public health, contemporary medicine is gradually reintegrating the use of complementary therapeutic methods. Music therapy is a non-medical intervention that is particularly suited to pain problems. The therapeutic use of music is an economical, practical and safe method. Many clinical studies show that this activity promotes a significant decrease in pain. The ability of passive listening to music to reduce the perception of pain has been called "music-induced analgesia". The neuro-psycho-physiological mechanisms that underlie this phenomenon remain poorly understood. One hypothesis, still discussed, proposes that listening to music would stimulate, directly or indirectly, endogenous mechanisms of modulation of pain, stemming from the brainstem. In individuals undergoing nociceptive tonic stimulation, the specific neuronal activation induced by listening to music demonstrates the involvement of inhibitory descending pathways. A measurement of pain control mechanisms would account for the impact of music on central awareness.

The purpose of this research is therefore to study the neuromodulatory effect of music on the sensory component of pain. The activation of pain control systems, through music, would pave the way for rehabilitation prospects for patients with a deficit of these controls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 65
* Subjects informed of the constraints of the study and having given their written consent.
* Subjects benefiting from a social security scheme.

Exclusion Criteria:

* Subjects under 18 and over 65
* Subjects who have previously participated in a pain study involving the induced pain test.
* Subjects with serious psychiatric disorders.
* Subjects with a diagnosis of acute or chronic pain.
* Subjects who have been taking antalgic substances for less than a week.
* Subjects with progressive disease not stabilized by medical treatment.
* Women in menstruation.
* Pregnant women.
* Subjects with a score greater than 10 for the Depressive Dimension on Hospital Anxiety and Depression Scale (HADS)
* Subjects with an anxiety score "state" higher than anxiety "traits" on the Spielberger condition state / traits anxiety inventory (STAI)
* Subjects with a score of 32 or higher on the Catastrophe Rating Scale (PCS-CF)
* Non-cooperating person.
* Person under legal protection
* Subjects not benefiting from a social security scheme
* Refusal of participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of Visual Analogue scale (VAS) | 20 minutes
  Visual Analogue Scale (VAS) measured at 2 minutes of stimulation during the temporal summation phase, starting from a basic VAS calibrated at 50/100.
  Pain is assessed continuously throughout this test using a computerized analog visual scale.

SECONDARY OUTCOMES:
Average VAS of the subject over the period P1 | 2 minutes
  The period P1 represents the first stimulation or the first time summation test. It is a tonic pain test by applying the thermode. The average VAS will be measured during this period.
  Pain is assessed continuously throughout this test using a computerized analog visual scale.
Average VAS of the subject over the period P2 | 2 minutes
  The period P2 represents the second stimulation or activation of the DNIC (Diffuse Nociceptive Inhibitive Control). This is the induction of cold thermal nociceptive stimulation (CPT : cold pressor test). The average VAS will be measured during this period.
  Pain is assessed continuously throughout this test using a computerized analog visual scale.
Average VAS of the subject over the period P3 | 2 minutes
  The period P3 represents the third stimulation or the second time summation test. This is the second tonic pain test by applying the thermode.The average VAS will be measured during this period.
  Pain is assessed continuously throughout this test using a computerized analog visual scale.
Evaluation of numerical scale | 20 minutes
  Numerical scale (overall numerical scale over the period) will be measured for each stimulation period (P1, P2, P3).
  This scale assesses pain and is graded from 0 (no pain) to 100 (maximum pain imaginable).
Difference in average VAS P1-P3 | 20 minutes
  The difference in average VAS between period P1 and period P3 will be calculated.
  Pain is assessed continuously throughout this test using a computerized analog visual scale.
Difference in Pressure Pain Threshold (PPT) before and after the procedure | 1 hour and 30 minutes
  The difference in Pressure Pain Threshold (PPT) will be measured before and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gildas L'Heveder, MD, Study Director — Brest University Hospital in France; Céline Bodere, MD, Principal Investigator — Brest University Hospital in France
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.